CLINICAL TRIAL: NCT00774579
Title: Growth Hormone Replacement in Adults With Growth Hormone Deficiency (GHD) - The Effect on Liver Fat.
Brief Title: The Effect of Growth Hormone Replacement on Liver Fat
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GHD1
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2009-12

CONDITIONS: Growth Hormone, Recombinant; Fatty Liver
Keywords: growth hormone; growth hormone deficiency; liver fat; liver steatosis; growth hormone replacement
MeSH Terms: conditions — Fatty Liver; Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, serum, leucocytes, 24-hour urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with growth hormone (GH) deficiency starting GH replacement.
- 2: Patients with growth hormone (GH) deficiency not starting GH replacement.

SUMMARY:
We will examine a cohort of growth hormone deficient adults starting growth hormone (GH) replacement. The purpose of this study is to determine whether GH replacement reduces the fat content of the liver.

To compare the results we will include growth hormone deficient patients who do not start GH replacement as controls.

DETAILED DESCRIPTION:
Adults with untreated growth hormone deficiency (GHD), a condition mostly due to pituitary disease, often show metabolic features similar to those described in the 'metabolic syndrome'. Growth hormone (GH) replacement has been shown to reverse many of these unfavorable changes, with a particular evident reduction of visceral fat. In recent years, a strong correlation between fat accumulation in the liver and features of the metabolic syndrome (particularly visceral fat) has been identified, and 'fatty liver' is now being referred as the hepatic feature of the 'metabolic syndrome'. The effect of GH replacement on liver fat, however, has never been systematically studied.

We will assess 15 patients with GHD before and 6 months after starting GH replacement. We will also assess 15 control patients with GHD but who don't go on GH replacement for various reasons.

Liver fat will be assessed using MR spectroscopy. Changes in liver fat will be correlated to changes in insulin sensitivity and changes in various inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* 20-70 years of age
* Growth hormone deficiency, with (cohort 1) or without (cohort 2) planned growth hormone (GH) replacement
* clinically stable

Exclusion Criteria:

* known hepatic disease
* Acromegaly
* Diabetes mellitus
* growth hormone replacement within the last 12 months
* cushing's disease, if not cured for at least 12 months
* any contraindication to MR studies as set out in the MR safety questionnaire

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the endocrine clinics of Imperial College Healthcare NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabian A Meienberg, Dr, Study Chair — Imperial College London; Stephen Robinson, Dr, Study Chair — Imperial College London; Jeremy Cox, Dr, Study Chair — Imperial College London; Ian Godsland, Dr, Study Chair — Imperial College London; Jimmy Bell, Dr, Study Chair — Imperial College London; Desmond G Johnston, Prof, Principal Investigator — Imperial College London; Simon Taylor-Robinson, Prof, Study Chair — Imperial College London; Emma Hatfield, Dr, Study Chair — Imperial College London; Michael Yee, Dr, Study Chair — Imperial College London
Locations (1):
- Endocrinology & Metabolic Medicine, Imperial College, London, United Kingdom

REFERENCES:
- [Derived] Meienberg F, Yee M, Johnston D, Cox J, Robinson S, Bell JD, Thomas EL, Taylor-Robinson SD, Godsland I. Liver fat in adults with GH deficiency: comparison to matched controls and the effect of GH replacement. Clin Endocrinol (Oxf). 2016 Jul;85(1):76-84. doi: 10.1111/cen.13042. Epub 2016 Mar 22. PMID 26895949

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2008 and April 2009 adult hypopituitary patients with untreated GHD were identified and recruited at the endocrine clinics of Imperial College Healthcare NHS Trust.
Groups:
- GH Replacement: Patients with growth hormone (GH) deficiency starting GH replacement.
- Control: Patients with growth hormone (GH) deficiency not starting GH replacement.
Period: Overall Study
Arm/Group | GH Replacement | Control
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GH Replacement | Control | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (8) | 52 (9) | 52 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Intrahepatocellular Lipid (IHCL) Content
Description: IHCL content determined by proton magnetic resonance spectroscopy (1H MRS).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | GH Replacement | Control
Number analyzed (Participants) | 9 | 9
% change from baseline | -0.63 (4.53) | 0.11 (1.46)
Statistical Analysis 1: Comparison: GH Replacement vs Control; Test type: Superiority; p = 0.6, t-test, 2 sided

2. Secondary Outcome: Total Adipose Tissue
Description: total adipose tissue assessed by MRI scan
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | GH Replacement | Control
Number analyzed (Participants) | 9 | 9
kg | -1.8 (3.2) | 0.24 (2.28)
Statistical Analysis 1: Comparison: GH Replacement vs Control; Test type: Superiority; p = 0.1, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | GH Replacement | Control
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes